CLINICAL TRIAL: NCT04794140
Title: A Randomized Controlled, Blinded, Prospective Clinical Study Evaluating the Effect of Endoscopic Ultrasound-guided Fine-needle Biopsy With Different Number of Passes on the Success Rate of Primary Cell Culture of Pancreatic Cancer
Brief Title: A Clinical Study to Evaluated Which Number of Passes of EUS-FNB is Better for Culturing Primary Cells of PDAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2021EUS-001
Record Dates: First submitted 2021-03-01; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- one pass group (Experimental): We use the endoscopic ultrasound-guided fine-needle biopsy (EUS-FNB) wet suction technique to procure the specimens, and use the sample obtained from a single pass for primary cell culture. EUS-FNB wet suction technique refer from Tong T, et al. J Gastroenterol Hepatol. 2020;10.1111/jgh.15371.
  Interventions: Procedure: different number of passes
- two passes group (Experimental): We use the endoscopic ultrasound-guided fine-needle biopsy (EUS-FNB) wet suction technique to procure the specimens, and use the sample obtained from two passes for primary cell culture. EUS-FNB wet suction technique refer from Tong T, et al. J Gastroenterol Hepatol. 2020;10.1111/jgh.15371.
  Interventions: Procedure: different number of passes

INTERVENTIONS:
Procedure: different number of passes — Each patient's operation process is the same, that is, after obtaining enough specimens for diagnosis by endoscopic ultrasound-guided fine-needle biopsy (EUS-FNB) wet suction technique, additional three passes are performed. One of which is randomly selected as the one pass group, and the other two passes automatically as the two pass group. Please refer to the literature for EUS-FNB wet technique (Tong T, et al. J Gastroenterol Hepatol. 2020;10.1111/jgh.15371.)

SUMMARY:
The Aim of this study is to investigate the amount of tissue required for the successful culture of primary cells from human-derived pancreatic ductal adenocarcinoma which obtained by endoscopic ultrasound-guided fine-needle biopsy wet suction technique

DETAILED DESCRIPTION:
Pancreatic cancer is one of the malignant tumors with the highest mortality rate in the world, with a 5-year survival rate of only 7.2%-9%. Because some patients are resistant to multiple chemotherapy drugs, and there are differences in drug sensitivity between individuals, the current pancreatic ductal adenocarcinoma (PDAC) chemotherapy effect is not satisfactory. In order to improve the efficacy of chemotherapy and achieve precise treatment, it is important to establish an accurate and individualized PDAC research model.

Because most of patients with PDAC have developed to advanced stage at the time of diagnosis, it is not suitable for surgery. That limits our ability to obtain tumor cells seriously. With the development of endoscopic ultrasound-guided fine-needle biopsy (EUS-FNB) technique, it can be used not only to diagnose diseases, but also to provide specimens for molecular analysis and create valuable preclinical disease research models, so as to guide the selection of the most appropriate individualized treatment. EUS-FNB can obtain lesions without any treatment. Therefore, the preclinical disease research model established by EUS-FNB is more representative of the original tumor.

However, compared with surgical specimens, the specimens obtained by EUS-FNB are smaller in size, which may affect the successful construction of research models in vitro. Therefore, the investigators plan to use EUS-FNB wet suction technique, a modified specimen acquisition method, to obtain PDAC tissue, and use it for primary cell culture, to explore the amount of tissue required for the successful cultivation of human-derived pancreatic cancer primary cells, so as to provide a prerequisite for the successful establishment of human-derived preclinical disease research model.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age≥18
2. Imaging examination (US, MRI, CT or PET-CT) of patients confirmed pancreatic lesions, and considered the possibility of PDAC, EUS-FNB was needed for auxiliary diagnosis
3. No chemotherapy, including neoadjuvant chemotherapy, postoperative adjuvant chemotherapy and palliative chemotherapy, has been performed on patients
4. Agree to attend this study and signed informed consent

Exclusion Criteria:

1. Poor physical condition, including but not limited to hemoglobin ≤ 8.0g/dl, severe cardiopulmonary insufficiency, etc
2. Coagulation dysfunction (platelet count < 50 × 1012, international standardized ratio > 1.5), or inability to discontinue anticoagulation therapy
3. High risk for deep sedation
4. Acute pancreatitis in the previous 2 weeks
5. Pregnancy or lactation
6. Any diseases leading to unreliable follow-up
7. Absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Differences in the success rate of culturing primary cells | About 6 weeks after operation
  Differences in the success rate of pancreatic cancer primary cells (P1) and culture to the third generation (P3) between the two groups.
The difference in the representation to the original tumor between the two groups of primary cells | About 8 weeks after operation
  Through Western Blot and PCR methods to detect the representativeness of primary cells to the primary tumor. If the patient underwent surgery later, hematoxylin-eosin staining and/or immunohistochemistry were added to compare the histological morphology with the original tumor.

SECONDARY OUTCOMES:
The relationship between the success rate of primary cell culture and some tumor characteristics | About 6 weeks after operation
  Statistical methods such as chi-square test are used to analyze whether the success rate of primary cell culture is related to the tumor size, degree of differentiation, clinical stage, and the length of macroscopic visible core tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyan Wang, M.D., Principal Investigator — The Third Xiangya Hospital, Central South University
Locations (1):
- The Third Xiangya Hospital, Central South University,, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No